CLINICAL TRIAL: NCT00571467
Title: An Open Label, Sequential, Dose Escalation, Repeat-dose Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of PRTX-100 in Adult Patients With Chronic Idiopathic Thrombocytopenic Purpura (ITP)
Brief Title: Phase I Safety and Tolerability Study of Staphylococcal Protein A in Adult Patients With Chronic ITP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to recruitment not meeting expectations.
Sponsor: Protalex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRTX-100A-201
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Idiopathic Thrombocytopenic Purpura (ITP)
Keywords: Autoimmune Diseases; Bleeding Disorders; Blood and Blood Disorders
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Autoimmune Diseases; Hemostatic Disorders; Hematologic Diseases | interventions — Staphylococcal Protein A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRTX-100 (Staphylococcal protein A) (Experimental): Cohort 1: 0.075 mcg/kg
  Cohort 2: 0.15 mcg/kg
  Cohort 3: 0.30 mcg/kg
  Interventions: Drug: PRTX-100 (Staphylococcal protein A)

INTERVENTIONS:
Drug: PRTX-100 (Staphylococcal protein A) — 4 weekly IV (in the vein) doses of 1 of the 3 following PRTX-100 dose levels:
  * Cohort 1: 0.075 mcg/kg
  * Cohort 2: 0.15 mcg/kg
  * Cohort 3: 0.30 mcg/kg
  Other Names: PRTX-100

SUMMARY:
The primary purpose of this study is to evaluate the safety of multiple doses of Staphylococcal protein A (PRTX-100) in adult patients with Idiopathic Thrombocytopenia Purpura (ITP). The pharmacokinetics, immunogenicity and pharmacodynamics will also be studied.

Patients will be enrolled into 1 of 3 dose groups and receive 4 weekly IV doses of PRTX-100. A Safety Monitoring Committee will review safety data through Day 28 for the first 5 patients in a dose group before escalation to the next higher dose level. Patients will be followed for 8 weeks after dosing for safety, PK, immunogenicity and effect on platelet count(pharmacodynamics).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic ITP > 4 months
* Mean platelet count <50 x 10^9/L for patients not receiving corticosteroids; or mean platelet count >=50 x 10^9/L for patients receiving stable dose of corticosteroids

Exclusion Criteria:

* Splenectomy within 45 days of screening
* Rituximab within 6 months prior to screening
* Cyclophosphamide, vincristine, or any other non-monoclonal antibody treatment for ITP within 3 months prior to screening
* IVIG, WinRho or other anti-RhD within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the overall safety of PRTX-100 during the 3 month study duration | 3 months

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of multiple doses of PRTX-100 | over the first 35 days
Explore immunogenicity of multiple doses of PRTX-10 | 3 months
Evaluate treatment effect on platelet count | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Bernton, MD, Study Director — Protalex, Inc.
Locations (7):
- Australia (6):
  - Canberra Hospital, Garran, Australian Capital Territory
  - St. George Hospital, Sydney, New South Wales
  - Royal Brisbane, Brisbane, Queensland
  - Monash Medical Centre, Melbourne, Victoria
  - Freemantle Hospital, Fremantle, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Middlemore Hospital, Otahuhu, Auckland, New Zealand